CLINICAL TRIAL: NCT05264519
Title: The Effect of Foot Bath on Premenstrual Syndrome, Sleep Quality and Quality of Life Among University Students With Premenstrual Syndrome
Brief Title: The Effect of Foot Bath on PMS, Sleep and Quality of Life Among University Students With PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hüsne YÜCESOY (Other)
Responsible Party: Sponsor-Investigator, Hüsne YÜCESOY, PROF. DR., Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HY1
Record Dates: First submitted 2021-11-22; First posted 2022-03-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Nursing; Foot Bath; Sleep Quality; Life Quality
MeSH Terms: conditions — Premenstrual Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): foot bath intervention
  Interventions: Other: foot bath intervention
- control (No Intervention): follow-up

INTERVENTIONS:
Other: foot bath intervention — Students in this group will have their feet soaked in water with a temperature of 38-42 degrees for 20 minutes, half an hour before bedtime.
  Arms: intervention

SUMMARY:
Premenstrual syndrome is a cyclical disorder characterized by physical and emotional symptoms that appear in the late luteal phase of the menstrual cycle and subside within a few days with the onset of menstruation. Non-pharmacological methods should be recommended first to women who experience PMS symptoms. For this purpose, it is planned to apply foot bath to university students with premenstrual syndrome.

The study was planned as a randomized controlled single-blind study. The universe of the research will be female students studying at Ordu University Faculty of Education in the 2021-2022 academic year. In the first stage of the study, female students who are 18 years of age and older and who voluntarily agree to participate in the research will be taken without making a sample selection. Considering the possibility of data loss during the research process, it was planned to work on 39 intervention and 39 control groups, including a total of 78 women In the collection of data; Personal Information Form, Premenstrual Syndrome Scale (PMSS), Pittsburgh Sleep Quality Index (PSQI), SF-36 Quality of Life Scale will be used. PSQI and SF-36 Quality of Life Scale will be applied to students in the intervention group. The foot bath will be applied for 3 months, starting 7-10 days before the menstrual cycle, that is, in the luteal phase of the menstrual cycle. Students will be asked to fill out the Footbath Monitoring Form in order to assess whether they have taken a footbath. Those who apply foot bath at least 7 times will be included in the study. In case of less than seven students, the student will be excluded from the research and the new student who meets the criteria will be included in the research. At the end of each cycle, PMSÖ, PSQI and SF-36 will be administered to the students by the researcher. When the students in the Control Group are determined, PSQI and SF-36 will be applied by the researcher, and then PMSÖ, PSQI and SF-36 will be applied at the end of each cycle.

DETAILED DESCRIPTION:
Premenstrual syndrome is a cyclical disorder characterized by physical and emotional symptoms that appear in the late luteal phase of the menstrual cycle and subside within a few days with the onset of menstruation. Although the etiology is not known precisely, many factors are thought to be effective. Premenstrual symptoms that occur in the second half of the menstrual cycle negatively affect the lives of many women. Pharmacological, non-pharmacological and surgical methods are used as treatment methods. Non-pharmacological methods should be recommended first to women who experience PMS symptoms. Non-pharmacological methods have advantages such as increasing the effectiveness of analgesic drugs, reducing the need for drugs, preventing the side effects of the drug and not bringing too much economic burden. For this purpose, it is planned to apply foot bath to university students with premenstrual syndrome. Although many studies have been conducted both in our country and abroad on university students' coping with PMS, no study has been found that investigates the effect of foot bathing on premenstrual syndrome severity, sleep quality and quality of life to cope with PMS.

The study was planned as a randomized controlled single-blind study. The universe of the research will be female students studying at Ordu University Faculty of Education in the 2021-2022 academic year. In the first stage of the study, female students who are 18 years of age and older and who voluntarily agree to participate in the research will be taken without making a sample selection. The number of students to be included in the intervention and control groups of the research will be determined according to the results of the power analysis in the G-Power 3.1.9.7 program. Considering the possibility of data loss during the research process, it was planned to work on 39 intervention and 39 control groups, including a total of 78 women, 10% of the calculated sample size. In the collection of data; Personal Information Form, Premenstrual Syndrome Scale (PMSS), Pittsburgh Sleep Quality Index (PSQI), SF-36 Quality of Life Scale will be used. PSQI and SF-36 Quality of Life Scale will be applied to students in the intervention (footbath) group by the researcher. Students will be given footbath practice training, which takes approximately 30-40 minutes. During the training, it will be shown how to apply foot bath. The foot bath will be applied for 3 months, starting 7-10 days before the menstrual cycle, that is, in the luteal phase of the menstrual cycle. The researcher will send a reminder message to the students every day for 7-10 days, starting 7-10 days before the period according to the previous menstrual period of the students. Students will be asked to fill out the Footbath Monitoring Form in order to assess whether they have taken a footbath. Those who apply foot bath at least 7 times will be included in the study. In case of less than seven students, the student will be excluded from the research and the new student who meets the criteria will be included in the research. At the end of each cycle, PMSÖ, PSQI and SF-36 will be administered to the students by the researcher. When the students in the Control Group are determined, PSQI and SF-36 will be applied by the researcher, and then PMSÖ, PSQI and SF-36 will be applied at the end of each cycle.

In this study, the effect of applying foot bath to university students with premenstrual syndrome on premenstrual syndrome symptoms, sleep quality and quality of life will be determined. It is thought that the low-cost, easy-to-apply foot bath will reduce symptoms and increase sleep quality and quality of life in women with PMS. As a result of the research, it will be possible to ensure that this application is among the other non-pharmacological methods used to cope with PMS and its use will become widespread. Thus, by increasing the sleep quality and quality of life of university students who are adversely affected by PMS symptoms, their school, work and social lives will be changed positively, and positive contributions will be made to their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older,
* Getting 111 points or more from the Premenstrual Syndrome Scale
* Being single
* Having a regular menstrual cycle for the last 6 months (every 21-35 days and no intermittent bleeding),
* Having a Body Mass Index (BMI) between 19-24.9,
* Not using cigarettes or alcohol,
* Not receiving medical treatment for PMS,
* Not receiving treatment for insomnia,

Exclusion Criteria:

* Having a psychiatric diagnosis
* Having a gynecological disease,
* Doing regular exercise,
* Using hormonal contraception (such as oral contraceptives and injections),

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | 20 minutes
  Students with PMS will be determined by applying the personal information form and PMSÖ to the students who accept to participate in the research. Then, PMSÖ, 1st, 2nd and 3rd cycles according to the groups. PMSÖ has nine sub-dimensions and consists of 44 questions. The lowest 44, the highest 220 points are taken from the scale. A high score indicates a greater intensity of PMS symptoms.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 20 minutes
  After the students with PMS are identified, an intervention and control group will be formed. PSQI will be applied to students in the intervention and control groups. Then, at the end of the 1st, 2nd and 3rd cycles, the Pittsburgh Sleep Quality Index will be applied.The PSQI score has a value between 0-21. A total PSQI score of 5 or less indicates good sleep quality, and a total of 6 and above indicates poor sleep quality.The PSQI score has a value between 0-21. A total PSQI score of 5 or less indicates good sleep quality, and a total of 6 and above indicates poor sleep quality.

OTHER OUTCOMES:
SF-36 Quality of Life Scale | 10 minutes
  After the students with PMS are identified, an intervention and control group will be formed. SF-36 Quality of Life Scale will be applied to students in the intervention and control groups. Then, at the end of the 1st, 2nd and 3rd cycles, the SF-36 Quality of Life Scale will be applied. From the SF-36 Quality of Life Scale, "0" indicates the lowest and "100" indicates the best level of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ordu Üniversitesi, Ordu, Altınordu
  - Ordu University, Ordu, Centre

IPD SHARING:
Plan to Share IPD: No